CLINICAL TRIAL: NCT05636540
Title: Evaluating in Vivo PARP-1 Expression With 18F-FluorThanatrace Positron Emission Tomography (PET/CT) in Patients With Pheochromocytoma and Paraganglioma
Brief Title: In Vivo PARP-1 Expression With 18F-FluorThanatrace PET/CT in Patients With Pheochromocytoma and Paraganglioma
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Heather Wachtel (Other)
Responsible Party: Sponsor-Investigator, Heather Wachtel, Assistant Professor of Surgery, Abramson Cancer Center at Penn Medicine
Organization: Abramson Cancer Center at Penn Medicine (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: UPCC 10322; 851463 (Other: University of Pennsylvania IRB)
Record Dates: First submitted 2022-10-20; First posted 2022-12-05 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Pheochromocytoma; Paraganglioma
MeSH Terms: conditions — Pheochromocytoma; Paraganglioma

STUDY DESIGN:
Intervention Model Description: This is a pilot observational study to determine the feasibility of [18F]FTT PET/CT to evaluate PARP-1 enzyme expression in pheochromocytoma/paraganglioma.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort A (Experimental): After undergoing screening assessments and verifying eligibility for study participation subjects will be scheduled to undergo a baseline experimental [18F]FTT PET/CT scan prior to surgery. Patients in Cohort A will undergo surgery with or without additional therapy.
  Interventions: Drug: [18F]FluorThanatrace ([18F]FTT)
- Cohort B (Experimental): After undergoing screening assessments and verifying eligibility for study participation subjects will be scheduled to undergo a baseline experimental [18F]FTT PET/CT scan prior to systemic therapy with radionuclide or chemotherapy. Up to 10 patients undergoing systemic therapy may undergo a second (optional) scan that will be performed approximately 1-21 days after therapy has started. The second scan is obtained to evaluate whether the initiation of systemic therapy alters [18F]FTT uptake. As this is a pilot study, only a limited number of patients are sought for the second scan.
  Interventions: Drug: [18F]FluorThanatrace ([18F]FTT)

INTERVENTIONS:
Drug: [18F]FluorThanatrace ([18F]FTT) — A pre-treatment 18F-FluorThanatrace ([18F]FTT) positron emission tomography/computed tomography (PET/CT) scan will be done prior to surgery or systemic therapy.

SUMMARY:
This study will enroll up to 30 evaluable patients with pheochromocytoma or paraganglioma who are undergoing surgical or systemic treatment.

A pre-treatment 18F-FluorThanatrace ([18F]FTT) positron emission tomography/computed tomography (PET/CT) scan will be done prior to surgery or systemic therapy.

PET/CT imaging will be used to evaluate PARP-1 expression in sites of pheochromocytoma or paraganglioma using the investigational radiotracer [18F]FTT. This is an observational study in that [18F]FTT PET/CT will not be used to direct treatment decisions. While patients and referring physicians will not be blinded to the [18F]FTT PET/CT results, treatment decisions will be made by the treating physicians based upon clinical criteria.

DETAILED DESCRIPTION:
Up to 30 patients who will undergo approximately 60 minutes of dynamic scanning head to thigh starting at approximately the same time as the injection, this will be followed by a second head to thigh scan [starting at approximately 90 minutes post injection. PET/CT imaging sessions will include an injection of ≤ 12 mCi of [18F]FTT intravenously (approximate range for most studies is anticipated to be 8-12 mCi).

If surgery is performed according to standard of care tissue will be processed for both clinical and research use, if the subject has consented for use of tissue. Data will be collected to evaluate uptake of [18F]FTT in pheochromocytoma and paraganglioma and compare with PARP-1 activity and other experimental assays in tissue from biopsy and surgery, when available.

All evaluable patients may undergo surgery or systemic therapy following the [18F]FTT PET/CT scan. Up to 10 patients undergoing systemic therapy may undergo a second (optional) scan that will be performed approximately 1-21 days after therapy has started. The second scan is obtained to evaluate whether the initiation of systemic therapy alters [18F]FTT uptake. As this is a pilot study, only a limited number of patients are sought for the second scan.

ELIGIBILITY:
Inclusion Criteria:

1. Participants will be ≥ 18 years of age.
2. Clinical diagnosis of pheochromocytoma or paraganglioma based on biochemical and imaging studies At least one lesion identified on standard of care imaging (e.g. CT, MRI, FDG or 68-Gallium dotatate, other PET/CT or MIBG).
3. Standard of care germline genetic testing performed for clinical purposes or participant's consent for germline genetic testing for research purposes.
4. Participants must be informed of the investigational nature of this study and be willing to provide written informed consent and participate in this study in accordance with institutional and federal guidelines prior to study-specific procedures.

Exclusion Criteria:

1. Inability to tolerate imaging procedures in the opinion of an investigator or treating physician.
2. Females who are pregnant or breastfeeding will not be eligible for this study; a urine pregnancy test will be performed in women of child-bearing potential prior to FTT injection.
3. Any current medical condition, illness, or disorder as assessed by medical record review and/or self-reported that is considered by a physician investigator to be a condition that could compromise participant safety or successful participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Standard uptake value (SUV)measurement - [F18]FTT | Baseline
  Qualitative measure SUV of [18F]FTT in phenochromocytoma/paraganlioma region (categories: positive, negative or mixed)
Maximum standard uptake value (SUV)measurement - [F18]FTT | Baseline
  Measure of maximum SUV of [18F}FTT in primary lesion region
Mean Standard uptake value (SUV)measurement - [F18]FTT | Baseline
  Measure of mean SUV of [18F}FTT in primary lesion region
Peak Standard uptake value (SUV)measurement - [F18]FTT | Baseline
  Measure of peak SUV of [18F}FTT in primary lesion region
Standard uptake value (SUV)measurement - [F18]FTT | Follow-Up (1-21 days post therapy)
  Qualitative measure SUV of [18F]FTT in phenochromocytoma/paraganlioma region (categories: positive, negative or mixed)
Maximum standard uptake value (SUV)measurement - [F18]FTT | Follow-Up (1-21 days post therapy)
  Measure of maximum SUV of [18F}FTT in primary lesion region
Mean Standard uptake value (SUV)measurement - [F18]FTT | Follow-Up (1-21 days post therapy)
  Measure of mean SUV of [18F}FTT in primary lesion region
Peak Standard uptake value (SUV)measurement - [F18]FTT | Follow-Up (1-21 days post therapy)
  Measure of peak SUV of [18F}FTT in primary lesion region

OTHER OUTCOMES:
Progression free survival (PFS) | From first day of treatment (PARP and/or ADT) to first documented disease progression or death due to any cause, assessed up to 10 years.
  Time from initial participation in study to disease progression or death from any cause,

CONTACTS AND LOCATIONS:
Overall Officials: Heather Wachtel, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No